CLINICAL TRIAL: NCT07365228
Title: OPEN SPACE AND CLOSED YEARS
Acronym: OS&CY
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Goran Kuvacic (Other)
Responsible Party: Sponsor-Investigator, Goran Kuvacic, Assistant Professor, University of Split
Organization: University of Split (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Open space and closed years; IP-UNIST-23_OPZG (Other Grant/Funding Number: Ministry of Science, Education and Youth of the Republic of Croatia)
Record Dates: First submitted 2025-12-21; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Physical Fitness; Health Literacy; Lipid Profile; Body Composition; Physical Literacy
Keywords: physical fitness; health status; postmenopausal women

STUDY DESIGN:
Intervention Model Description: Experimental (treatment group) vs. Control (non-treated group)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Evaluation (Experimental): Participants in the intervention
  Interventions: Behavioral: Physical exercising

INTERVENTIONS:
Behavioral: Physical exercising — Participants will be involved in regular physical exercising in public space

SUMMARY:
The primary objective of this project is to examine the effects of a specific multicomponent physical activity program (MPAP), conducted in an outdoor setting, on the health and functional-motor status (HFMS) of women over the age of 60. Additionally, the study will investigate the influence of sociodemographic factors (SDF), physical literacy (PL), and health literacy (HL) on the baseline HFMS and the subsequent changes resulting from the KTP.

Study Methodology

The program participants will consist of older women (>60 years; n=60) whose current HFMS allows for participation in the exercise protocol. They will be divided into two groups:

Experimental Group: Will participate in the MPAP.

Control Group: Will not participate in the MPAP.

The exercise intervention (MPAP) will include a combination of aerobic activities, strength exercises, balance, and flexibility. It will be conducted two to three times per week across two three-month cycles, separated by a three-month break.

Data Collection and Environment Assessments: Sociodemographic factors, physical literacy, and health literacy will be measured at the start of the study. A series of HFMS indicators will be recorded before and after each exercise cycle.

Setting: The MPAP will be performed outdoors in a public park.

Project Significance Beyond analyzing the direct effects of the exercise program and the correlations between the measured variables, this project will contribute to a deeper understanding of the importance of the natural environment in implementing goal-oriented physical activity for the elderly population.

DETAILED DESCRIPTION:
The primary objective of this project is to examine the effects of a specific multicomponent physical activity program (MPAP), conducted in an outdoor setting, on the health and functional-motor status (HFMS) of women over the age of 60. Additionally, the study will investigate the influence of sociodemographic factors (SDF), physical literacy (PL), and health literacy (HL) on the baseline HFMS and the subsequent changes resulting from the KTP.

Study Methodology

The program participants will consist of older women (>60 years; n=60) whose current HFMS allows for participation in the exercise protocol. They will be divided into two groups:

Experimental Group: Will participate in the MPAP.

Control Group: Will not participate in the MPAP.

The exercise intervention (MPAP) will include a combination of aerobic activities, strength exercises, balance, and flexibility. It will be conducted two to three times per week across two three-month cycles, separated by a three-month break.

Data Collection and Environment Assessments: Sociodemographic factors, physical literacy, and health literacy will be measured at the start of the study. A series of HFMS indicators will be recorded before and after each exercise cycle.

Setting: The MPAP will be performed outdoors in a public park.

Project Significance Beyond analyzing the direct effects of the exercise program and the correlations between the measured variables, this project will contribute to a deeper understanding of the importance of the natural environment in implementing goal-oriented physical activity for the elderly population.

ELIGIBILITY:
Inclusion Criteria:

* physical fitness status which allows active participation in the physical exercising program organized as a tretment

Exclusion Criteria:

* health conditions not allowing the participation in treatment program

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2029-06-01 (Estimated)

PRIMARY OUTCOMES:
Fitness status - dynamic balance | 3 months
  Measured by Biodex balance system on the basis of standardized protocol
Fitness status - static balance | 3 monts
  Measured by Biodex balance system using the standardized protocol
Lipid profile | 3 months
  Tryglicerides, LDL Cholesterol, HDL Cholesterol, Total Cholesterol (measured by POC testing device)
Health literacy | 3 months
  Health literacy evidenced via HLS19-Q12

SECONDARY OUTCOMES:
Body composition - skeletal muscle mass | 3 months
  Measured by Tanita measurement scale
Body composition - body fat | 3 months
  Measured by Tanita scale

OTHER OUTCOMES:
Physical literacy | 3 months
  Evidenced by PPLQ

IPD SHARING:
Plan to Share IPD: Undecided
Anonymity issues